CLINICAL TRIAL: NCT04524832
Title: A Randomised Trial Investigating Steady State Semaglutide Exposure of 25 and 50 mg of Oral Semaglutide in Different Formulations in Healthy Subjects
Brief Title: Research Study Comparing New Tablets of Semaglutide in New Doses, in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4633; U1111-1242-2643 (Other: World Health Organization (WHO); 2019-004157-80 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2020-08-21; First posted 2020-08-24 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Semaglutide D 50 mg (Experimental): Participants will receive once daily semaglutide D formulation tablets in a dose escalating manner for 16 weeks: 2.4 mg (week 1-2), 5.6 mg (week 3-4), 11.2 mg (week 5-8), 25 mg (week 9-12) and 50 mg (week 13-16)
  Interventions: Drug: Oral semaglutide
- Semaglutide C 50 mg (Experimental): Participants will receive once daily semaglutide C formulation tablets in a dose escalating manner for 16 weeks: 2.4 mg (week 1-2), 5.6 mg (week 3-4), 11.2 mg (week 5-8), 25 mg (week 9-12) and 50 mg (week 13-16)
  Interventions: Drug: Oral semaglutide
- 2 x Semaglutide C 25 mg (Experimental): Participants will receive once daily semaglutide C formulation tablets in a dose escalating manner for 16 weeks: 2.4 mg (week 1-2), 5.6 mg (week 3-4), 11.2 mg (week 5-8), 25 mg (week 9-12) and 2 x 25 mg (week 13-16)
  Interventions: Drug: Oral semaglutide
- Semaglutide E 50 mg (Experimental): Participants will receive once daily semaglutide tablets in a dose escalating manner for 16 weeks: A) Semaglutide C formulation: 2.4 mg (week 1-2), 5.6 mg (week 3-4) and 11.2 mg (week 5-8). B) Semaglutide E formulation: 25 mg (week 9-12) and 50 mg (week 13-16)
  Interventions: Drug: Oral semaglutide
- Semaglutide F 50 mg (Experimental): Participants will receive once daily semaglutide F formulation tablets in a dose escalating manner for 16 weeks: 2.4 mg (week 1-2), 5.6 mg (week 3-4), 11.2 mg (week 5-8), 25 mg (week 9-12) and 50 mg (week 13-16)
  Interventions: Drug: Oral semaglutide

INTERVENTIONS:
Drug: Oral semaglutide — Participants will receive once daily semaglutide tablets (oral administration) in a dose escalating manner for 16 weeks

SUMMARY:
In this study a known investigational medicinal product called semaglutide will be tested in four different tablet versions. In addition to semaglutide, the different tablet versions C, D, E and F contain different helping agents in different amounts. All tablet versions have a helping agent called SNAC. All tablet versions are tested for the treatment of type 2 diabetes. Recently the European Medicines Agency approved semaglutide in tablet form and currently, tablets in the doses 3 mg, 7 mg and 14 mg can be prescribed in some countries. The main aim of this study is to test oral semaglutide doses of 25 mg and 50 mg. These are higher dosages of oral semaglutide than can be prescribed today. With the 50 mg dose, we expect the amount of semaglutide in the blood to be higher than what has been tested before. Further aims of this study are to find an optimal version for the semaglutide tablets, and to examine the safety and tolerability of the different tablet versions. For this purpose, the amount of semaglutide in the blood will be measured after taking different semaglutide tablets, in different doses. The version of the tablet participants will receive (i.e. the treatment arm participants will be assigned to) is decided by chance.

In treatment periods 1 and 2 participants will receive one tablet daily over 2 weeks for each period. For treatment periods 3 to 5 participants will receive one tablet daily over 4 weeks for each period (participants may get 2 tablets per day in treatment period 5). This means that treatment will take 16 weeks in total. The tablets should be taken in the morning together with no more than half a glass of water (120 mL), after an overnight fast of at least 6 hours (no food or drinks). Water is also not allowed from 2 hours before dosing. After dosing participants must wait 30-35 minutes before they eat or drink. At home, participants must take their breakfast 30-45 minutes after dosing.

No oral medication (which are taken by mouth) can be taken from 2 hours before and until 30 minutes after each dosing with semaglutide. The study can last for up to 24 weeks for each participant. This includes a screening period (up to 3 weeks), a treatment period (16 weeks) and a follow-up visit (5 weeks after the last dosing). Participants will have 11 clinic visits with the study doctor. Some of the visits include overnight stays. Participants will have blood tests at every visit. Participants must be healthy and have a body mass index (BMI) between 21.0 and 29.9 kg/m^2 For women: Women cannot take part in this study if they are pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-64 years (both inclusive) at the time of signing informed consent.
* Body mass index between 21.0 kg/m^2 and 29.9 kg/m^2 (both inclusive).
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Glycated haemoglobin (HbA1c) greater than or equal to 6.5 % (48 mmol/mol) at screening.
* Use of tobacco and nicotine products, defined as any of the below:1) Smoking more than 5 cigarettes or the equivalent per day.2) Not willing to refrain from smoking and use of nicotine substitute products during the inpatient periods.
* Presence of clinically significant gastrointestinal disorders or symptoms of gastrointestinal disorders potentially affecting absorption of drugs or nutrients, as judged by the investigator.
* History (as declared by participant) of major surgical procedures involving the stomach potentially affecting absorption of trial products (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery).
* Personal or first degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma (as declared by participant).
* Presence or history (as declared by participant) of pancreatitis (acute or chronic).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 290 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Area under the semaglutide plasma concentration - time curve during a dosing interval at steady state (AUC0-24h,sema,SS) | From 0 to 24 hours after the last dosing of oral semaglutide 25 mg on visit 8, day 84
  nmol*h/L
Area under the semaglutide plasma concentration-time curve during a dosing interval at steady state (AUC0-24h,sema,SS) | From 0 to 24 hours after the last dosing of oral semaglutide 50 mg on visit 10, day 112
  nmol*h/L

SECONDARY OUTCOMES:
Area under the semaglutide plasma concentration-time curve during a dosing interval at steady state (AUC0-24h,sema,SS) | From 0 to 24 hours after the last dosing of oral semaglutide 11.2 mg on visit 6, day 56.
  nmol*h/L
Maximum semaglutide plasma concentration at steady state (Cmax,sema,SS) | From 0 to 24 hours after the last dosing of oral semaglutide 11.2 mg on visit 6, day 56
  nmol/L
Maximum semaglutide plasma concentration at steady state (Cmax,sema,SS) | From 0 to 24 hours after the last dosing of oral semaglutide 25 mg on visit 8, day 84
  nmol/L
Maximum semaglutide plasma concentration at steady state (Cmax,sema,SS) | From 0 to 24 hours after the last dosing of oral semaglutide 50 mg on visit 10, day 112
  nmol/L
Time to maximum semaglutide plasma contraction at steady state (tmax,sema,SS) | From 0 to 24 hours after the last dosing of oral semaglutide 25 mg on visit 8, day 84
  hour
Time to maximum semaglutide plasma contraction at steady state (tmax,sema,SS) | From 0 to 24 hours after the last dosing of oral semaglutide 50 mg on visit 10, day 112
  hour
Number of treatment-emergent adverse events | From the time of first dosing (visit 2, day 1) until completion of the follow-up visit (visit 11, day 149)
  Count
Change in pulse | From baseline (visit 2, day 1) to end of treatment (visit 10, day 113)
  Beats/minute
Change in blood pressure | From baseline (visit 2, day 1) to end of treatment (visit 10, day 113)
  mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure 1452, Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com